CLINICAL TRIAL: NCT06273228
Title: An Online Parenting Intervention for Families Affected by Substance Misuse in Pediatric Primary Care
Brief Title: Parenting Young Children in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000788; P50DA048756 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Parenting; Parent-Child Relations; Substance Use Disorders; Stress; Depression; Anxiety; Parenting Self-efficacy; Pediatrics
Keywords: Parenting Intervention; Family Check-Up
MeSH Terms: conditions — Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parents will be recruited in pediatric primary care settings and will be assessed at baseline and at a 3-month follow-up. Parents will receive the intervention between baseline and follow-up. Nine parents will be randomly selected for an additional follow-up interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent participants (Experimental): Parents receive access to the FCU Online website and telehealth coaching/ support provided by a trained mental health provider. The FCU Online website includes a brief 5-minute assessment, feedback on parents' responses, and online tools to support parenting in areas that were identified as challenges by the assessment. These tools include animated videos, parenting tips, and interactives to help practice parenting skills. Telehealth coaching will focus on Wellness and Self-Care, Parenting and Substance Use, Positive Parenting, Proactive Parenting, and Supervision and Limit Setting.
  Interventions: Behavioral: Family Check-Up Online

INTERVENTIONS:
Behavioral: Family Check-Up Online — This intervention includes access to the Family Check-Up Online website and telehealth coaching provided by trained mental health providers.

SUMMARY:
In this study, investigators will partner with pediatric primary care providers to recruit parent participants, then evaluate feasibility and acceptability by systematically assessing parents' engagement with the FCU Online app. Engagement data from the app includes time spent in app overall and in each module, activities completed, and which modules were accessed. Investigators will also administer a consumer satisfaction survey, which will ask parents to report on their perceptions of the app (e.g., helpfulness, useability, and effects on parenting). To assess engagement in telehealth coaching sessions, investigators will use the following variables: number of telehealth sessions completed, length of session, content of sessions, and coaches' ratings of participant engagement in the session and barriers to using the app. Coaches will also rate participant engagement on a 3-point scale from "low" to "high." Lastly, investigators will conduct qualitative interviews with a sub-sample of participants to solicit additional feedback on the acceptability of the FCU Online, focusing particularly on the perception of acceptability within an integrated primary care context and stigma associated with endorsing substance use in this setting.

DETAILED DESCRIPTION:
Research suggests that one in eight children in the U.S. currently lives with a parent with a substance use disorder. Parents who misuse substances are at increased risk of using harsh and other negative parenting practices with their young children, who are more likely to face challenges with emotional and behavioral regulation and subsequently misuse substances themselves. There is thus an urgent need for evidence-based interventions to promote positive parenting skills in parents who misuse substances. Interventions must be convenient, non-stigmatizing, and accessible to parents with problematic substance use, who frequently face barriers to engaging with healthcare systems. Pediatric primary care is an ideal setting to offer a brief intervention for maladaptive parenting behaviors associated with parental substance use, as the vast majority of children under 5 access pediatric primary care at least annually and parents generally report high levels of trust in their child's pediatrician.

The Family Check-Up (FCU) Online app, which was created specifically to promote positive parenting skills in parents with past or current substance misuse, is ideal for delivery to parents with pre-school age children in a pediatric primary care setting as it is brief, convenient, and delivered in a self-directed format that parents favor. The main objective of this pilot study is to test the feasibility and acceptability of the FCU-Online, a brief, app-based parenting intervention, for parents reporting lifetime problematic substance use in a pediatric primary care setting.

In this study, investigators will partner with pediatric primary care providers to recruit parent participants, then evaluate feasibility and acceptability by systematically assessing parents' engagement with the FCU Online app. Engagement data from the app includes time spent in app overall and in each module, activities completed, and which modules were accessed. Investigators will also administer a consumer satisfaction survey, which will ask parents to report on their perceptions of the app (e.g., helpfulness, useability, and effects on parenting). To assess engagement in telehealth coaching sessions, investigators will use the following variables: number of telehealth sessions completed, length of session, content of sessions, and coaches' ratings of participant engagement in the session and barriers to using the app. Coaches will also rate participant engagement on a 3-point scale from "low" to "high." Lastly, investigators will conduct qualitative interviews with a sub-sample of participants to solicit additional feedback on the acceptability of the FCU Online, focusing particularly on the perception of acceptability within an integrated primary care context and stigma associated with endorsing substance use in this setting.

A second aim of this study is to assess pediatric healthcare providers' perceptions and attitudes regarding the fit of the FCU Online with their practice settings as well as potential barriers to implementation. Through semi-structured focus groups and qualitative interviews with pediatric healthcare providers, investigators will assess provider- and practice-level factors that may facilitate or impede the implementation of the FCU Online in pediatric primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Must be a parent of a child between the ages of 10 months and 5 years that lives in the parent's home at least 50% of the time;
* Must be over the age of 18;
* Must speak English fluently;
* Must have a smart phone with text messaging capability and access to email;
* Must endorse "yes" on at least one of the five following screening questions addressing lifetime family substance misuse: 1) participant has ever drunk alcohol or used drugs more than they meant to, 2) participant has ever participated in treatment for substance use, 3) participant has ever felt they wanted or needed to cut down on their drinking or drug use, 4) participant ever ever lived with someone who had a problem with drinking or using drugs, including prescription drugs, and 5) a family member's drinking or drug use ever impacted the participant's child. Note: Items 1, 3, and 5 were adapted from the Family Questions section of the Survey of Well-Being of Young Children (SWYC) screening form, which has been recommended by the American Academy of Pediatrics for use as a screening tool in pediatric primary care settings. Adaptations made reflect lifetime family substance misuse instead of family substance misuse in the past year. Item 2 was added to include parents in substance use treatment, and item 4 was adapted from the Adverse Childhood Experience Questionnaire for Adults to further reflect family substance use.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
change from baseline in parenting skills | Time Frame: baseline, 3 months
  Parenting skills will be measured with the Parenting Young Children Questionnaire (PARYC). Scores range from 1-7; a higher score indicates more positive parenting.
change from baseline in parenting efficacy | baseline, 3 months
  Parenting self-efficacy will be measured with the Behavioral Self-Efficacy subscale (PAREFF) of the Parenting Tasks Checklist. Scores range from 1-5; a higher score indicates greater parenting efficacy.
change from baseline in parent executive functioning | baseline, 3 months
  Parent executive functioning will be measured with the Behavior Rating Index of Executive Function (BRIEF). Scores range from 1-3; a higher score indicates greater difficulty with executive function.
change from baseline in child social-emotional behavior | baseline, 3 months
  Child social-emotional behavior will be measured with the Brief Infant-Toddler Social-Emotional Assessment (BITSEA). Scores range from 1-3; a higher score indicates more positive child social-emotional behavior.
change from baseline in family conflict | baseline, 3 months
  Family conflict will be measured with the Family Conflict Scale. Scores range from 1-7; a higher score indicates a higher frequency of family conflict.
change from baseline in parental depression | baseline, 3 months
  Parental depression will be measured with the Patient Health Questionnaire-9 (PHQ-9). Scores range from 0-3; a higher score indicates greater depression.
change from baseline in parental anxiety | baseline, 3 months
  Parental anxiety will be measured with the General Anxiety Disorder-7 (GAD-7). Scores range from 0-3; a higher score indicates greater anxiety.
change from baseline in parental stress | baseline, 3 months
  Parental stress will be measured with the Perceived Stress Scale. Scores range from 0-56; a higher score indicates high perceived stress.
change from baseline in parental impact of negative life events | baseline, 3 months
  The impact of negative life events will be measured with the life events subscale of the Parent Self-Check (PARSC). Scores range from 1-5; a higher score indicates greater impact of negative life events.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hails, PhD, Principal Investigator — University of Oregon
Locations (1):
- Prevention Science Institute, University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT06273228/ICF_001.pdf